CLINICAL TRIAL: NCT00589888
Title: Free Fatty Acids-Induced Hypertension and Endothelial Dysfunction in Obese Subjects
Brief Title: FFA-Induced Hypertension and Endothelial Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, MD, Professor of Medicine, Emory University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB00041116; IRB 668-2006 (Other: Other)
Record Dates: First submitted 2007-12-28; First posted 2008-01-10 (Estimated); Results first posted 2014-07-09 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Endothelial Dysfunction; Hypertension
Keywords: hypertension; metabolic syndrome; vascular reactivity; Elevated blood pressure; lipid toxicity
MeSH Terms: conditions — Hypertension; Metabolic Syndrome | interventions — soybean oil, phospholipid emulsion; Saline Solution; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Intralipid 20%@ 20cc/hour (Active Comparator): Intralipid 20% IV infusion at 20cc/hour
  Interventions: Drug: Intralipid 20% @ 20cc/hour
- Intralipid 20% @ 40cc/hour (Active Comparator): Intralipid 20% IV infusion at 40cc/hour
  Interventions: Drug: Intralipid 20%@ 40cc/hour
- Normal Saline infusion @ 40cc/hour (Placebo Comparator): Normal Saline continuous IV infusion at 40cc/hour for 8 hours
  Interventions: Drug: Normal Saline
- 32-gram oral fat load (Active Comparator): 32-gram oral fat load once
  Interventions: Dietary Supplement: 32-gram oral fat load
- 64-gram oral fat load (Active Comparator): 64-gram oral fat load once
  Interventions: Dietary Supplement: 64-gram oral fat load

INTERVENTIONS:
Drug: Intralipid 20% @ 20cc/hour — In this arm subjects received Intralipid 20% Intravenous IV continuous infusion at 20cc/hour for 8 hours. The 20% intralipid solution is a long-chain triglyceride emulsion composed of 50% polyunsaturated fatty acids, 26% monounsaturated fatty acids, and 19% saturated fatty acids. During the intralipid infusion studies, subjects remained fasting
  Other Names: 20% i.v. fat emulsion
  Arms: Intralipid 20%@ 20cc/hour
Drug: Intralipid 20%@ 40cc/hour — In this arm subjects received Intralipid 20% IV continuous infusion at 40cc/hour for 8 hours. In this arm subjects will receive Intralipid 20% Intravenous IV continuous infusion at 20cc/hour for 8 hours. The 20% intralipid solution is a long-chain triglyceride emulsion composed of 50% polyunsaturated fatty acids, 26% monounsaturated fatty acids, and 19% saturated fatty acids. During the intralipid infusion studies, subjects remained fasting.
  Other Names: 20% i.v. fat emulsion
  Arms: Intralipid 20% @ 40cc/hour
Drug: Normal Saline — In this arm subjects received 0.9% Normal Saline continuous IV infusion at 40/cc for 8 hours.
  Other Names: 0.9% Sodium Chloride
  Arms: Normal Saline infusion @ 40cc/hour
Dietary Supplement: 32-gram oral fat load — In this arm subjects received oral liquid fat load prepared by the General Clinical Research Center (GCRC) at baseline and every 2 hours for 6 hours. Participants received fat with Free Fatty Acids (FFA) composed of 33% polyunsaturated fatty acids, 34% monounsaturated fatty acids, and 22% saturated fatty acids. The oral fat load in either low or high dose was given in four equally divided doses at 0, 2, 4, and 6 h.
  Arms: 32-gram oral fat load
Dietary Supplement: 64-gram oral fat load — In this arm subjects received 60-gram oral fat load intake at baseline and every 2 hours for 6 hours prepared by the General Clinical Research Center (GCRC). Participants received fat with Free Fatty Acids (FFA) composed of 33% polyunsaturated fatty acids, 34% monounsaturated fatty acids, and 22% saturated fatty acids. The oral fat load in either low or high dose was given in four equally divided doses at 0, 2, 4, and 6 h.
  Arms: 64-gram oral fat load

SUMMARY:
The study is a prospective open label study to examine the effects of oral and intravenous fat load on blood pressure, endothelial function, sympathetic activity, and oxidative stress in obese healthy subjects. Subjects will receive either 8-hour of intravenous or oral fat loads in either low or high doses or normal saline in random order. Blood samples are drawn and vitals are measured before and after the infusions. Endothelial function and plasma glucose and lipid levels are measured to study the effects.

DETAILED DESCRIPTION:
Insulin resistance has been implicated as the central mechanism in the development of several cardiovascular risk factors including hypertension, diabetes, lipid disorders, and coagulation disorders. Recent evidence suggests that increased levels of a circulation fat (free fatty acids or FFAs) are a leading candidate causing insulin resistance. Our preliminary studies in indicate that, in addition to insulin resistance, the infusion of Intralipid and heparin to increase FFAs resulted in a significant rise in systolic and diastolic blood pressure, impaired endothelial (vascular) function, and increased inflammatory markers in obese African Americans with and without diabetes. The effects of FFA on insulin action are well established; however, the blood pressure and vascular effects of FFAs infusion in obese subjects have not been fully investigated. We hypothesize that observed changes in blood pressure are the result of acute endothelial dysfunction, and/or increased activation of the autonomic nervous system. No previous studies have attempted to determine a dose response effect of increasing FFA on blood pressure. In addition, it is not know if increased FFAs by repeated oral fat load results in similar blood pressure than intravenous lipid infusion. Accordingly, we propose: 1) a systematic evaluation of the effects of increasing FFA levels on blood pressure and endothelial (vascular) function, and 2) determine the effects of comparable increases in FFA concentration via intravenous infusion of Intralipid or by repeated oral fat load on blood pressure, insulin resistance and endothelial dysfunction in obese subjects.

A group of obese normotensive subjects will be admitted to the Grady Clinical Research Center or to the Outpatient Research Unit in the Grady Diabetes Clinic on five occasions. In four of these admissions, research subjects will receive an 8-hour intravenous infusion, in random order, of increasing Intralipid concentration (10 ml, 20 ml, 40 ml per hour) or normal saline (40 ml per hour). During the final admission, research subjects will receive an oral liquid fat diet every 2 hours for 8-hours. The effect of increased FFAs on blood pressure and endothelial (vascular) function via intravenous infusion and via oral fat load therapy will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the ages of 18 and 65 years.
* Definition: obese = BMI ≥ 30 kg/m2
* Blood pressure < 140/80 mm Hg and no prior history of hypertension

Exclusion Criteria:

* History of hypertension or previous history of antihypertensive drug therapy.
* Current tobacco use
* Fasting triglyceride levels > 250 mg/dL during the stabilization period.
* Liver disease (ALT 2.5x > upper limit of normal), or other significant medical or surgical illness, including myocardial ischemia, congestive heart failure, liver failure, and infectious processes.
* Serum creatinine ≥1.5 mg/dL for males, or ≥ 1.4 mg/dL for females.
* History of drug or alcohol abuse within the last 5 years.
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
* Female subjects are pregnant or breast feeding at time of enrollment into the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-08; Primary Completion 2008-04 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University SOM/GCRC
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Result] Gosmanov AR, Smiley DD, Robalino G, Siquiera J, Khan B, Le NA, Patel RS, Quyyumi AA, Peng L, Kitabchi AE, Umpierrez GE. Effects of oral and intravenous fat load on blood pressure, endothelial function, sympathetic activity, and oxidative stress in obese healthy subjects. Am J Physiol Endocrinol Metab. 2010 Dec;299(6):E953-8. doi: 10.1152/ajpendo.00469.2010. Epub 2010 Oct 5. PMID 20923960

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For this study, same 13 subjects were admitted to the General Clinical Research Center at Grady Memorial Hospital in random order on five different occasions to receive either 8-h iv or oral fat loads in either low or high doses or normal saline.
Groups:
- Normal Saline @ 40cc/Hour: Normal Saline continuous IV infusion at 40cc/hour for 8 hours
  0.9% Normal Saline: 0.9% Normal Saline continuous IV infusion at 40/cc for 8 hours
- Intralipid 20% @ 20cc/hr: Intralipid 20% IV infusion at 20cc/hour
  Intralipid 20%: Intralipid 20% IV continuous infusion at 20cc/hour for 8 hours
- Intralipid 20% @ 40cc/Hour: Intralipid 20% IV infusion at 40cc/hour
  Intralipid 20%: Intralipid 20% IV continuous infusion at 40cc/hour for 8 hours
- 32-gram Oral Fat Load: 32-gram oral fat load
  32-gram oral fat load: oral liquid fat load prepared by the GCRC every 2 hours for 8 hours.
- 64-gram Oral Fat Load: 64-gram oral fat load
  64-gram oral fat load: 60-gram oral fat load intake every 2 hours for 8 hours
Period: Normal Saline @ 40cc/Hour
Arm/Group | Normal Saline @ 40cc/Hour | Intralipid 20% @ 20cc/hr | Intralipid 20% @ 40cc/Hour | 32-gram Oral Fat Load | 64-gram Oral Fat Load
Started | 13 (the same 13 patients did each of the 5 arms at 5 different visits) | 0 | 0 | 0 | 0
Completed | 13 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Intralipid 20% @ 20cc/hr
Arm/Group | Normal Saline @ 40cc/Hour | Intralipid 20% @ 20cc/hr | Intralipid 20% @ 40cc/Hour | 32-gram Oral Fat Load | 64-gram Oral Fat Load
Started | 0 (the same 13 patients did each of the 5 arms at 5 different visits) | 13 | 0 | 0 | 0
Completed | 0 | 13 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Intralipid 20% @ 40cc/Hour
Arm/Group | Normal Saline @ 40cc/Hour | Intralipid 20% @ 20cc/hr | Intralipid 20% @ 40cc/Hour | 32-gram Oral Fat Load | 64-gram Oral Fat Load
Started | 0 | 0 (the same 13 patients did each of the 5 arms at 5 different visits) | 13 (the same 13 patients did each of the 5 arms at 5 different visits) | 0 | 0
Completed | 0 | 0 | 13 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: 32-gram Oral Fat Load
Arm/Group | Normal Saline @ 40cc/Hour | Intralipid 20% @ 20cc/hr | Intralipid 20% @ 40cc/Hour | 32-gram Oral Fat Load | 64-gram Oral Fat Load
Started | 0 | 0 | 0 (the same 13 patients did each of the 5 arms at 5 different visits) | 13 (the same 13 patients did each of the 5 arms at 5 different visits) | 0
Completed | 0 | 0 | 0 | 13 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: 64-gram Oral Fat Load
Arm/Group | Normal Saline @ 40cc/Hour | Intralipid 20% @ 20cc/hr | Intralipid 20% @ 40cc/Hour | 32-gram Oral Fat Load | 64-gram Oral Fat Load
Started | 0 | 0 | 0 | 0 (the same 13 patients did each of the 5 arms at 5 different visits) | 13 (the same 13 patients did each of the 5 arms at 5 different visits)
Completed | 0 | 0 | 0 | 0 | 13
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: obese, healthy subjects. The same 13 participants received the interventions in random order on different occasions
Groups:
- All Study Participants: All participants received all 5 arms in random order:
  1. 0.9% Normal Saline continuous IV infusion at 40/cc for 8 hours
  2. Intralipid 20% @ 20cc/hr for 8 hours
  3. Intralipid 20% @ 40cc/Hr for 8 hours
  4. 32-gram Oral Fat Load every 2 hours for 8 hours.
  5. 64-gram Oral Fat Load every 2 hours for 8 hours.
Arm/Group | All Study Participants
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Baseline Flow-mediated dilatation (FMD) of Brachial Artery [Mean (Standard Deviation); unit: percentage] — FMD was assessed as a measurement of endothelial function. Ultrasound images of the brachial artery were obtained at baseline under standardized conditions and 60 s after induction of reactive hyperemia by 5-min cuff occlusion of the forearm. All images were digitized online, and arterial diameters were measured with customized software by individuals blinded to the clinical and laboratory status of the subjects. Flow-mediated dilatation (FMD) was expressed as the percentage increase in diameter from baseline. Itis measured in percentage
  percentage | 9.4 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure to After Completing an 8-hour Normal Saline Infusion in Obese Normotensive Subjects.
Description: To study the effects of high dose oral fat load on systolic blood pressure (SBP) in healthy obese subjects, subject's baseline SBP is compared to SBP after the infusion. Blood Pressure (BP) was measured with a manual cuff in triplicate on admission when patient was in Supine position. The Blood pressure was measured at admission and at end of the fat load. The BP from the admission are compared to BP after the fat load. A normal systolic blood pressure is lower than 120 mmHg; elevated blood pressure if the systolic reading is 120-129 mmHg. A level above 140 mmHg is considered hypertension.
Time Frame: Baseline and at the end of the 8-hours
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Normal Saline @ 40cc/Hour
Number analyzed (Participants) | 13
mmHg | 13 (17)

2. Primary Outcome: Change in Systolic Blood Pressure From Baseline to After Completing an 8-hour 20% Intralipid @ 20cc/hr Infusion in Obese Normotensive Subjects.
Description: To study the effects of low dose intravenous (IV) fat infusion on systolic blood pressure (SBP) in healthy obese subjects, subject's baseline SBP is compared to SBP after the infusion. Blood Pressure (BP) was measured with a manual cuff in triplicate on admission when patient was in Supine position. The Blood pressure was measured at admission and at every 2 hours till the end of infusion. The BP from the admission are compared to BP after the infusion.A normal systolic blood pressure is lower than 120 mmHg; elevated blood pressure if the systolic reading is 120-129 mmHg. A level above 140 mmHg is considered hypertension.
Time Frame: Baseline and at the end of the 8-hours
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Intralipid @ 20cc/Hour: Intralipid continuous IV infusion at 20cc/hour for 8 hours
Arm/Group | Intralipid @ 20cc/Hour
Number analyzed (Participants) | 13
mmHg | 14 (10)

3. Primary Outcome: Changes in Systolic Blood Pressure From Baseline to After Completing an 8-hour 20% Intralipid @ 40cc/hr Infusion in Obese Normotensive Subjects
Description: To study the effects of high dose intravenous (IV) fat infusion on systolic blood pressure (SBP) in healthy obese subjects, subject's baseline SBP is compared to SBP after the infusion. Blood Pressure (BP) was measured with a manual cuff in triplicate on admission when patient was in Supine position. The Blood pressure was measured at admission and at every 2 hours till the end of infusion. The BP from the admission are compared to BP after the infusion. A normal systolic blood pressure is lower than 120 mmHg; elevated blood pressure if the systolic reading is 120-129 mmHg. A level above 140 mmHg is considered hypertension.
Time Frame: Baseline and at the end of the 8-hours
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Intralipid @ 40cc/Hour for 8 Hours: Intralipid continuous IV infusion at 40cc/hour for 8 hours
Arm/Group | Intralipid @ 40cc/Hour for 8 Hours
Number analyzed (Participants) | 13
mmHg | 12 (9)

4. Primary Outcome: Change in Systolic Blood Pressure From Baseline to After Completing an Oral 32-gram Fat Load in Obese Normotensive Subjects.
Description: To study the effects of oral low dose fat load on systolic blood pressure (SBP) in healthy obese subjects, subject's baseline SBP is compared to SBP after the infusion. Blood Pressure (BP) was measured with a manual cuff in triplicate on admission when patient was in Supine position.The Blood pressure was measured at admission and at end of the fat load. The BP from the admission are compared to BP after the fat load. A normal systolic blood pressure is lower than 120 mmHg; elevated blood pressure if the systolic reading is 120-129 mmHg. A level above 140 mmHg is considered hypertension.
Time Frame: Baseline and at the end of the 8-hours
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Oral 32-gram Fat Load: For the low (32 g fat) oral fat load studies, participants received fat with FFA composed of 33% polyunsaturated fatty acids, 34% monounsaturated fatty acids, and 22% saturated fatty acids. The oral fat load in either low or high dose was given in four equally divided doses at 0, 2, 4, and 6 h.
Arm/Group | Oral 32-gram Fat Load
Number analyzed (Participants) | 13
mmHg | 13 (17)

5. Primary Outcome: Changes in Systolic Blood Pressure From Baseline to After Completing an Oral 64-gram Fat Load in Obese Normotensive Subjects
Description: as for outcome 1
Time Frame: at the end of the 8 hours
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Oral 64-gram Fat Load: For the high (64 g fat) oral fat load studies, participants received fat with FFA composed of 33% polyunsaturated fatty acids, 34% monounsaturated fatty acids, and 22% saturated fatty acids. The oral fat load in either low or high dose was given in four equally divided doses at 0, 2, 4, and 6 h.
Arm/Group | Oral 64-gram Fat Load
Number analyzed (Participants) | 13
mmHg | 11 (11)

6. Secondary Outcome: Change in Flow-mediated Dilation (FMD) of Endothelium-dependent Brachial Artery From Baseline to After Completing a Specific Intervention in Obese Normotensive Subjects.
Description: Endothelium-dependent brachial artery dilatation was assessed as a measurement of endothelial function using established methodology. Briefly, ultrasound images of the brachial artery were obtained at baseline under standardized conditions and 60 s after induction of reactive hyperemia by 5-min cuff occlusion of the forearm. Image landmarks as well as surface markers were utilized to ensure anatomic consistency between serial imaging studies. All images were digitized online, and arterial diameters were measured with customized software by individuals blinded to the clinical and laboratory status of the subjects. Flow-mediated dilatation (FMD) was expressed as the percentage increase in diameter from baseline. It is measured in percentage.
Time Frame: Baseline and at the end of the 8-hours
Measure: Mean (Standard Deviation); unit: percentage of FMD
Arm/Group | Intralipid 20%@ 20cc/Hour | Intralipid 20% @ 40cc/Hour | Normal Saline Infusion @ 40cc/Hour | 32-gram Oral Fat Load | 64-gram Oral Fat Load
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 13
percentage of FMD | 3.8 (2.1) | 4.1 (3.1) | 0.3 (0.1) | 3.8 (1.8) | 5 (2.5)

7. Secondary Outcome: Change in Blood Glucose Levels From Baseline to 6-8 Hours After Intervention Among Obese Healthy Subjects
Description: The blood glucose level is the amount of glucose present in the blood of humans. Many factors affect a person's blood sugar level. The body's homeostatic mechanism of blood sugar regulation (known as glucose homeostasis), when operating normally, restores the blood sugar level to a narrow range of about 4.4 to 6.1 mmol/L (79 to 110 mg/dL) (as measured by a fasting blood glucose test). The study aims to study the effects of these interventions on blood glucose levels among obese healthy subjects.
Time Frame: Baseline and at the end of the 8-hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intralipid 20%@ 20cc/Hour | Intralipid 20% @ 40cc/Hour | Normal Saline Infusion @ 40cc/Hour | 32-gram Oral Fat Load | 64-gram Oral Fat Load
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 13
mg/dL
  baseline blood glucose level | 93.9 (4.4) | 92.3 (9.2) | 91.5 (8.5) | 91.5 (6.4) | 87.1 (4.0)
  After intervention blood glucose level | 84.2 (5.7) | 86.1 (8.1) | 81.7 (7.2) | 87.8 (7.8) | 87.8 (10.3)

8. Secondary Outcome: Change in C-peptide Concentration Levels From Baseline to After Specific Intervention Among the Healthy Obese Subjects
Description: C-peptide is a peptide composed of 31 amino acids. It is released from the pancreatic beta-cells during cleavage of insulin from proinsulin. It is mainly excreted by the kidney, and its half-life is 3-4 times longer than that of insulin. The reference range of C-peptide is 0. 8-3 ng/ml. The C-peptide test is a tool to monitor and treat diabetes. It shows how well your body makes insulin, which moves sugar (or "glucose") from your blood into your cells.
Time Frame: baseline and after 8 hours after admission
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Intralipid 20%@ 20cc/Hour | Intralipid 20% @ 40cc/Hour | Normal Saline Infusion @ 40cc/Hour | 32-gram Oral Fat Load | 64-gram Oral Fat Load
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 13
ng/ml
  baseline C- Peptide | 1.64 (0.84) | 2.06 (0.69) | 1.95 (0.87) | 2.02 (0.59) | 2.5 (0.41)
  After intervention C- Peptide level | 2.1 (1.08) | 2.05 (0.62) | 1.49 (0.63) | 2.51 (0.78) | 2.49 (1.03)

9. Secondary Outcome: Change in Blood Insulin Levels From Baseline to After Intervention Among the Normal Obese Subjects
Description: Insulin is an anabolic hormone that promotes glucose uptake, glycogenesis, lipogenesis, and protein synthesis of skeletal muscle and fat tissue through the tyrosine kinase receptor pathway. In addition, insulin is the most important factor in the regulation of plasma glucose homeostasis, as it counteracts glucagon and other catabolic hormones like epinephrine, glucocorticoid, and growth hormone. Normal fasting insulin levels is < 25 milli-International unit/litre
Time Frame: Baseline and at the end of the 8-hours
Population: the same 13 subjects underwent different interventions in random order on different occasions
Measure: Mean (Standard Deviation); unit: milli-International unit /Litre
Arm/Group | Intralipid 20%@ 20cc/Hour | Intralipid 20% @ 40cc/Hour | Normal Saline Infusion @ 40cc/Hour | 32-gram Oral Fat Load | 64-gram Oral Fat Load
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 13
milli-International unit /Litre
  baseline blood insulin | 8.5 (7.1) | 9.2 (4.5) | 8.8 (5) | 7.8 (4.1) | 9.1 (2.7)
  After intervention blood insulin level | 8.6 (5.7) | 9.1 (4.4) | 5.2 (3.5) | 11.5 (6) | 12.9 (9.4)

ADVERSE EVENTS:
Time Frame: From baseline (time of admission) to completing the intervention that is 8 hours.
Arm/Group | Normal Saline @ 40cc/Hour | Intralipid 20% @ 20cc/hr | Intralipid 20% @ 40cc/Hour | 32-gram Oral Fat Load | 64-gram Oral Fat Load
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/13 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 1/13 | 1/13 | 0/13 | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Saline @ 40cc/Hour (N=13) | Intralipid 20% @ 20cc/hr (N=13) | Intralipid 20% @ 40cc/Hour (N=13) | 32-gram Oral Fat Load (N=13) | 64-gram Oral Fat Load (N=13)
venous irritation (Vascular disorders) | 0 | 1 | 1 | 0 | 0 — temporary irritation of vein towards the end of the 8-hour infusion; no permanent sequelae or discontinuation
indigestion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 — temporary symptoms of reflux after ingesting the meal; no permanent sequelae or discontinuation

LIMITATIONS AND CAVEATS:
The study subjects were mostly African-Americans, precluding generalization of the findings to other ethnic groups. Study was of short duration, and the composition of oral fat load was not identical to the intralipid composition.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No